CLINICAL TRIAL: NCT04092166
Title: Impact of a Structured Cardiac Rehabilitation Program on Cardiorespiratory Fitness in Patients With Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Valley Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18.0090
Record Dates: First submitted 2019-07-03; First posted 2019-09-17 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled (No Intervention): Participants will have no intervention.
- Cardiac Rehab Exercise: Stationary Bike (Other): Participants will use a stationary bike machine that also engages the arms and use . This will be performed for 6 minutes, 3 times a week for a total of 8 weeks).
  Interventions: Other: Stationary Bike

INTERVENTIONS:
Other: Stationary Bike — Participants will use a stationary bike machine that also engages the arms and use . This will be performed for 6 minutes, 3 times a week for a total of 8 weeks).
  Arms: Cardiac Rehab Exercise: Stationary Bike

SUMMARY:
The objective of this study is to determine whether participation in an 8-week structured cardiac rehabilitation program can increase cardiorespiratory fitness in patients with atrial fibrillation.

DETAILED DESCRIPTION:
The study is a randomized, prospective single center study to assess the utility and efficacy of cardiac rehabilitation in patients with AF. All participants will receive the same medical care and standard baseline education which includes an hour long one on one session with a nutritionist.

Participants will also receive the guide book, Lifestyle Guide to Healing the Heart, at their baseline visit as part of their education

After obtaining informed consent to participate in the study and signing a consent form to participate in the Phase 3 cardiac rehabilitation program, participants will undergo a baseline assessment of their functional status using the functional capacity NuStep test. The NuStep test will be conducted at the Valley Hospital at baseline and after 8 weeks using the NuStep TRS 4000 machine - a stationary bike machine that also engages one's arms by pushing and pulling arm handles. Participants will sit in the NuStep machine and bike on level 4 (a low to moderate level) for 6 minutes, if possible. However, participants will be encouraged to step as quickly as possible during this time period. Participants will be asked about any discomfort before, during and after the test. The participant's METS are calculated directly by the machine based on the watts while exercising.

The degree of improvement of the participant's METS over the course of the 8-week program will produce a greater understanding of the effect of a structured cardiac rehabilitation program on cardiorespiratory fitness.

Following this baseline assessment, participants will then be randomized to undergo usual care or an 8-week (24-session) Phase 3 cardiac rehabilitation program at the Valley Health System Center for Health & Wellness in Mahwah. Eight weeks later, participants will undergo repeat assessment of functional status.

In addition, participants will be administered the Atrial Fibrillation Effect on Quality-of-life (AFEQT) survey at baseline, 6-months and 12-months later.

Patients will also undergo a 1-week Zio XT Holter monitor at the same time points (baseline, 6-months and 12-months). The Zio XT Holter monitor is a small, discreet comfortable patch that sticks on a participant's chest to test for any arrhythmias, such as AF duration and burden. The Zio XT Holter monitor will be available through commercial (HIPAA-compliant) remote monitoring portals and will not be stored locally in Valley Health System. However, in the future this may change and the Zio XT Holter monitor data will be stored as part of the participant's electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Individuals with paroxysmal or persistent AF
* Individuals with a BMI between 27 and 40

Exclusion Criteria:

* Inability to engage with a cardiac rehabilitation program
* Pregnant women
* If patient can perform exercise at a high intensity (6 METS or above), they will no longer be analyzed in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Will a cardiac rehab program increase cardiorespiratory fitness in Afib patients? | 1 year
  The primary endpoint of the study is to determine whether engagement with an 8-week, 24- session cardiac rehabilitation program can increase exercise capacity by 2 METS, a threshold that has previously been shown to improve patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, MD, Principal Investigator — The Valley Hospital
Locations (1):
- The Valley Hospital, Paramus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No